CLINICAL TRIAL: NCT02989753
Title: Pilot Study to Assess Effects of Two Herbal Dietary Supplements on Lipid Metabolism in Moderate Hypercholesterolemia and Hypertriglyceridemia
Brief Title: Effects of Two Herbal Dietary Supplements on Lipid Metabolism in Moderate Hypercholesterolemia and Hypertriglyceridemia
Acronym: Lipiback
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-A01178-43
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-05

CONDITIONS: Hypercholesterolemia; Hypertriglyceridemia
Keywords: Prevention
MeSH Terms: conditions — Hypercholesterolemia; Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): The comparative product is a placebo with the same characteristics of appearance and packaging as studied products and in which all ingredients are replaced by maltodextrin.
  Interventions: Dietary Supplement: Placebo
- VAL070-A (Experimental): Studied active product n°1, named VAL070-A, is a dietary supplement in shape of capsule. VAL070-A product contains 4 active plant extracts.
  Interventions: Dietary Supplement: VAL070-A
- VAL070-B (Experimental): Studied active product n°2, named VAL070-B, is a dietary supplement in shape of capsule. VAL070-B product contains 5 active plant extracts.
  Interventions: Dietary Supplement: VAL070-B

INTERVENTIONS:
Dietary Supplement: VAL070-A — After randomization (V1 visit), 8 capsules per day of VAL070-A during 12 weeks (from visit V1 to visit V2). They will consume 3 capsules at the beginning of their breakfast, 2 capsules at the beginning of their lunch and 3 capsules at the beginning of their dinner.
  Arms: VAL070-A
Dietary Supplement: VAL070-B — After randomization (V1 visit), 8 capsules per day of VAL070-B during 12 weeks (from visit V1 to visit V2). They will consume 3 capsules at the beginning of their breakfast, 2 capsules at the beginning of their lunch and 3 capsules at the beginning of their dinner.
  Arms: VAL070-B
Dietary Supplement: Placebo — After randomization (V1 visit), 8 capsules per day of placebo during 12 weeks (from visit V1 to visit V2). They will consume 3 capsules at the beginning of their breakfast, 2 capsules at the beginning of their lunch and 3 capsules at the beginning of their dinner.
  Arms: Placebo

SUMMARY:
This study is designed as a pilot study in order to estimate the effect of VAL070-A and VAL070-B products and their variability on LDL cholesterol and lipid metabolism since these data are still unknown for these products and in this specific population. Collected data will provide more reliable information which may be used to plan a subsequent larger main study.

DETAILED DESCRIPTION:
Main objective

The primary objective of the present trial is to assess the beneficial effect of VAL070-B compared to a placebo, on blood LDL cholesterol level in moderate hypercholesterolemic and hypertriglyceridemic subjects after 12 weeks of consumption.

Secondary objectives

Secondary objectives of the study are to assess the effects of VAL070-A and VAL070-B, compared to a placebo and to each other, in moderate hypercholesterolemic and hypertriglyceridemic subjects after 12 weeks if consumption through the following parameters:

* Blood level of LDL cholesterol (VAL070-A compared to placebo and VAL070-A compared to VAL070-B),
* Lipid profile: Blood levels of triglycerides, total cholesterol, HDL-cholesterol and non- HDL cholesterol,
* Glycaemia,
* Blood hsCRP,
* Fructosamine,
* Blood total free fatty acid levels,
* Anthropometrics assessed by body weight (BW), waist circumference (WC), hip circumference (HC) and waist to hip ratio (WHR).

Safety objectives

The following parameters, analyzed at baseline and after 12 weeks of consumption, participated to the safety objectives:

* Blood levels of urea and creatinine,
* Blood levels of GGT, AST and ALT,
* Complete blood count,
* Hemodynamic measurements: heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP),
* Adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years (limits included),
* BMI between 18.5 and 40 kg/m2 (limits included),
* For women: Non menopausal with the same reliable contraception since at least 3 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study (condom with spermicide gel and estrogen/progestin combination contraception accepted) or menopausal without or with hormone replacement therapy (estrogenic replacement therapy begun from less than 3 months excluded),
* Weight stable within ± 5 % in the last three months,
* Non smoking or with tobacco consumption < 20 cigarettes / day,
* Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme,
* Agree to be registered on the volunteers in biomedical research file.

After V1 biological analysis the subjects will be eligible to the study on the following criteria:

* Fasting blood LDLc level (using Friedewald estimation method) between 1.3 and 2.2 g/L (limits included with ± 2 % tolerated around),
* Fasting blood triglycerides level > 1.5 g/L,
* Blood TSH level between 0.27 and 4.2 μIU/mL (limits included).

Within 3 months following to the exit of the study for failure to comply to one or more of the inclusion criteria listed above, a re-screening could be performed.

Exclusion Criteria:

* Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal trouble or other metabolic disorder,
* Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease),
* With a history of ischemic cardiovascular event,
* Having undergone recent surgical procedure (less than 6 months),
* Suffering from an uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg),
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient,
* Pregnant or lactating women or intending to become pregnant within 3 months ahead,
* For women: pregnancy or breastfeeding finished since less than 6 months,
* Under cholesterol and/or lipid-lowering treatment (e.g. statins, fibrates, ezetimibe, bile acid sequestrants, niacin, etc.) or stopped less than 3 months before the V1 visit,
* Requiring a cholesterol lowering by immediate pharmacologic intervention according to the current recommendations (AFSSAPS, 2005),
* Under medication which could affect blood lipid parameters (e.g. long-term corticosteroid systemic drug, systemic antibodies, androgens or enzyme inducer, etc.) or stopped less than 3 months before the randomization (antihypertensive stable long-term treatment tolerated),
* Regular intake of dietary supplements or "functional foods" which are known to have an impact on lipid metabolism (e.g. rich in plant stanol or sterol like PRO-ACTIV or DANACOL products, red yeast rice, policosanol, capsules containing omega-3 fatty acids from fish oils, containing beta glucanes, konjac extract or cinnamon, etc.) or stopped less than 3 months before the V1 visit,
* Under treatment or dietary supplement which could significantly affect parameter(s) followed during the study according to the investigator or stopped in a too short period before the V1 visit,
* With significant change in food habits or in physical activity in the 3 months before the V1 visit or not agreeing to keep them unchanged throughout the study,
* With a current or planned in the next 3 months specific diet (hyper or hypocaloric, vegan, vegetarian...) or stopped less than 3 months before the study,
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator,
* Consuming more than 3 standard drinks of alcoholic beverage daily for men or 2 daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study,
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 10 hours of significant physical activity a week, walking excluded),
* Who made a blood donation in the 3 months before the V1 visit or intending to make it within 3 months ahead,
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency,

After V1 biological analysis the subjects will be considered as non eligible to the study on the following criteria:

* Fasting blood triglycerides > 4 g/L,
* Fasting glycaemia > 1.26 g/L
* Blood AST, ALT or GGT > 3xULN (Upper Limit of Normal),
* Blood urea > 12.11 mmol/L (value corresponding to 1.5xULN) or creatinine > 125 μmol/L,
* Blood hsCRP > 10 mg/L,
* Complete blood count with clinically significant abnormality according to the investigator.

Within 3 months following to the exit of the study for failure to comply to one or more of the exclusion criteria listed above, a re-screening could be performed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Comparison between VAL070-B and placebo on changes between V1 and V2 visits of the fasting blood LDL cholesterol | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g/L

SECONDARY OUTCOMES:
Comparison between VAL070-A and placebo on changes between V1 and V2 visits of the fasting blood LDL cholesterol | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g/L
Changes in fasting blood concentrations of triglycerides | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g/L
Changes in fasting blood concentrations of total cholesterol | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g/L
Changes in fasting blood concentrations of HDL cholesterol | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g/L
Changes in fasting blood concentrations of non-HDL cholesterol | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g/L
Changes in fasting blood concentrations of glucose | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in g/L
Changes in fasting blood concentrations of hsCRP | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in mg/L
Changes in fasting blood concentrations of fructosamine | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in µmol/L
Changes in fasting blood concentrations of total free fatty acid | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in mmol/L
Changes in body weight | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in kg
Changes in waist circumference | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in cm
Changes in hip circumference | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in cm
Changes in waist to hip ratio | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline)
Changes in fasting blood concentrations of urea | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in mmol/L
Changes in fasting blood concentrations of creatinine | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in µmol/L
Changes in fasting blood concentrations of AST (Aspartate aminotransferase) | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in µkat/L
Changes in fasting blood concentrations of ALT (Alanine aminotransferase) | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in µkat/L
Changes in fasting blood concentrations of GGT (Gamma glutamyltransferase) | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in µkat/L
Changes in complete blood count | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline)
Changes in heart rate | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in bpm
Changes in systolic blood pressure | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in mmHg
Changes in diastolic blood pressure | 12 weeks
  Defined as the difference V2 (12 weeks) - V1 (baseline) in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: David GENDRE, Dr, Principal Investigator — Biofortis Mérieux NutriSciences; Jean-Marie BARD, Dr-PhD, Study Chair — UFR des Sciences Pharmaceutiques et Biologiques, Nantes, France; Sébastien PELTIER, PhD, Study Director — Valbiotis
Locations (1):
- Biofortis Mérieux NutriSciences Clinical Investigation Center, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: Undecided